CLINICAL TRIAL: NCT07129109
Title: Assessing the Performance of 7-Day vs 1-Day Packaging for Small Quantity Lipid-Based Nutrient Supplements in Ghana (SQLNS:7Dv1D Comparison)
Brief Title: Assessing the Performance of 7-Day vs 1-Day Packaging for Small Quantity Lipid-Based Nutrient Supplements in Ghana (SQLNS:7D-1D Comparison)
Acronym: SQLNS:7Dv1D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of Ghana (Other); Edesia Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: SQLNS7
Record Dates: First submitted 2025-08-05; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Child Malnutrition
Keywords: Small-quantity lipid-based nutrient supplments (SQ-LNS); Ghana; Infant and young child feeding; Growth monitoring and promotion (GMP)
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SQ-LNS 1-day packaging first, followed by 7-day packaging (Active Comparator): SQ-LNS 1-day packaging first, followed by 7-day packaging
  Interventions: Dietary Supplement: small-quantity lipid-based nutrient supplements (SQ-LNS)
- SQ-LNS 7-day packaging first, followed by 1-day packaging (Experimental): SQ-LNS 7-day packaging first, followed by 1-day packaging
  Interventions: Dietary Supplement: small-quantity lipid-based nutrient supplements (SQ-LNS)

INTERVENTIONS:
Dietary Supplement: small-quantity lipid-based nutrient supplements (SQ-LNS) — All caregivers will receive 2 months of SQ-LNS in this cross-over design. Half of the participants will be randomized to receive the 7-day packaging first, and half will receive the 1-day packaging first.

SUMMARY:
This cluster-randomized crossover trial evaluates the impact of two different packaging formats for small-quantity lipid-based nutrient supplements (SQ-LNS) on adherence and acceptability among caregivers of young children in Northern Ghana. SQ-LNS are a proven intervention for reducing child malnutrition, but optimizing packaging formats may improve adherence and scalability.

Eight health facilities participating in growth monitoring services will each receive both formats: a 1-day sachet (20g daily) and a 7-day bulk container (140g weekly), with the order of delivery randomized. Each packaging format will be distributed for one month before cross-over. The primary outcomes are adherence (measured through caregiver self-report and sachet counts) and acceptability (assessed via caregiver interviews). Secondary outcomes include caregiver preference, ease of use, and qualitative insights into feeding practices, beliefs, and packaging usability.

This implementation research study uses a convergent mixed-methods design, integrating quantitative adherence and acceptability data with in-depth interviews and structured observations to inform real-world program implementation. Findings will guide policy and program decisions for integrating SQ-LNS into child health platforms in Ghana and other low-resource settings.

DETAILED DESCRIPTION:
Background and Rationale:

Small-quantity lipid-based nutrient supplements (SQ-LNS) have demonstrated effectiveness in reducing child undernutrition, including stunting, wasting, and anemia, particularly among children 6-24 months of age in low- and middle-income countries. Despite strong evidence, uptake and adherence in real-world settings remain suboptimal. Packaging format may influence how caregivers understand, use, and integrate SQ-LNS into daily routines.

This study, titled "Assessing the performance of 7-day vs 1-day packaging for Small Quantity Lipid-based Nutrient Supplements in Ghana," is designed to evaluate how packaging format influences adherence and acceptability when SQ-LNS are distributed through routine growth monitoring services in Northern Ghana.

Study Objectives:

Primary Objective: To compare adherence to SQ-LNS when delivered in 1-day sachets versus 7-day bulk packaging.

Secondary Objectives: To assess caregiver acceptability, preferences, ease of use, and perceptions of both packaging types; and to explore implementation facilitators and barriers to effective delivery and use of SQ-LNS within growth monitoring programs.

Study Design:

This is a cluster-randomized crossover trial embedded within routine child health services at eight health facilities. The trial follows a convergent mixed-methods implementation research design.

Clusters: Health facilities (n=8), each randomized to one of two packaging sequences.

Intervention: Each facility receives one packaging format for one month, then switches to the alternate format for another month.

Participants: Caregivers of children aged 6-24 months attending growth monitoring and promotion (GMP) services during the intervention periods.

Randomization:

Facilities are randomized to one of two sequences:

Sequence A: 1-day sachet → 7-day bulk Sequence B: 7-day bulk → 1-day sachet

Randomization is stratified by facility size or service volume (if available) to ensure balance.

Sample Size:

Based on prior service utilization data and expected recruitment rates, the study aims to enroll approximately 250 caregivers per facility per arm.

Outcomes:

Primary Outcomes:Adherence to SQ-LNS (measured by caregiver self-report, sachet count, and possibly biomarkers or stool colorant testing if available)

Secondary Outcomes:

Caregiver acceptability and preference (structured surveys and Likert scales) Usability and ease of administration Qualitative themes related to packaging, feeding practices, and caregiver experience (in-depth interviews and structured observations)

Data Collection:

Quantitative data will be collected through baseline and endline caregiver surveys, adherence logs, and observational checklists.

Qualitative data will be collected through purposive sampling of caregivers for in-depth interviews, as well as interviews with health workers and program implementers.

Analysis Plan:

Quantitative data will be analyzed using generalized linear mixed models to account for clustering and crossover design. Primary comparisons will assess differences in adherence between packaging formats. Qualitative data will be coded and analyzed thematically using a grounded theory approach.Convergence of quantitative and qualitative data will inform implementation recommendations.

Ethical Considerations:

The study will be submitted for IRB approval from received approval from Boston University and the University of Ghana. Written informed consent will be obtained from all participants. The study poses minimal risk and is embedded in routine health services.

Dissemination:

Findings will be shared with Ghana Health Service, implementing partners, and international stakeholders, and will be submitted for publication in peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child aged 6-24 months attending growth monitoring and promotion (GMP) services at one of the participating health facilities
* Willing and able to provide informed consent
* Plans to remain in the area for the duration of the study period
* Agrees to participate in surveys and/or interviews related to supplement use

Exclusion Criteria:

* Caregiver of a child with a diagnosed severe illness requiring hospitalization
* Caregiver under the age of 18

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Adherence | Measured twice per participant: at the end of the first 1-month phase and at the end of the second 1-month phase
  Adherence will be defined as the percentage of the 28-day dose of small quantity lipid-based nutrient supplements (SQ-LNS) consumed, measured using a triangulated approach that combines caregiver report with returned-sachet counts and residual-sachet weighing.

SECONDARY OUTCOMES:
Caregiver acceptability/usability | Measured twice per participant: at the end of the first 1-month phase and at the end of the second 1-month phase
  Caregiver acceptability/usability will be defined as a composite score (Likert-scaled) capturing acceptability, preference, usability, and ease of administration of the SQ-LNS packaging
Caregiver experience with SQ-LNS | At the end of each 1-month crossover period (following each intervention phase)
  Qualitative assessment of caregiver experience with SQ-LNS, including perceptions of packaging, feeding practices, and overall acceptability, collected through semi-structured interviews and analyzed using thematic content analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Eight health facilities in the Northern Region of Ghana (exact sites TBD), Tamale, Ghana

IPD SHARING:
Plan to Share IPD: No